CLINICAL TRIAL: NCT00293722
Title: Prospective Post Marketing Surveillance to Evaluate the Safety and Efficacy of Etanercept Under Usual Care Settings in Patients With Psoriatic Arthritis (PsA) Treated by Rheumatologists
Brief Title: Study Evaluating the Safety and Efficacy of Etanercept in Patients With Psoriatic Arthritis Treated by Rheumatologists
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A6-102064; B1801127
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Arthritis, Psoriatic; Psoriasis; Skin Diseases, Papulosquamous
Keywords: Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Skin Diseases, Papulosquamous; Arthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Psoriatic Arthritis
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — The patients will be treated in accordance with the requirements of the labelling of Enbrel® in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of etanercept under usual care settings in patients with PsA treated by rheumatologists.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriatic arthritis

Exclusion Criteria:

* Sepsis or risk for sepsis,
* Acute infection,
* Hypersensitivity against Etanercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients for whom the decision has already been made to initiate treatment with Enbrel® can be enrolled in this observational trial. These patients must have a proven diagnosis of Psoriatic Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 1308 (Actual)
Dates: Start 2006-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Toerwang-Samerberg, Germany

REFERENCES:
- [Derived] Behrens F, Meier L, Prinz JC, Jobst J, Lippe R, Loschmann PA, Lorenz HM. Simultaneous Response in Several Domains in Patients with Psoriatic Disease Treated with Etanercept as Monotherapy or in Combination with Conventional Synthetic Disease-modifying Antirheumatic Drugs. J Rheumatol. 2018 Jun;45(6):802-810. doi: 10.3899/jrheum.170932. Epub 2018 Apr 1. PMID 29606665
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A6-102064&StudyName=Study%20Evaluating%20the%20Safety%20and%20Efficacy%20of%20Etanercept%20in%20Patients%20with%20Psoriatic%20Arthritis%20Treated%20by%20Rheumatologists

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Psoriatic Arthritis: Participants with psoriatic arthritis treated by rheumatologist who received etanercept (Enbrel) as per local medical practice under conditions of routine daily use, were observed for 1 year.
Period: Overall Study
Arm/Group | Participants With Psoriatic Arthritis
Started | 1291
Completed | 864
Not Completed | 427
Not completed — Other | 427

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled in this study and had safety data available. Out of a total of 1285 participants included in the safety analysis set, data for baseline measure (age) was available only for 1274 participants.
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1285
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 708
  Male | 571
  Missing | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and Week 52 (end of the observation period) that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to Week 52
Population: Safety analysis set included all participants who were enrolled in this study and had safety data available.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1285
percentage of participants
  AEs | 38.1
  SAEs | 6.0

2. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Psoriasis at Week 52
Time Frame: Baseline, Week 52
Population: Efficacy analysis set included all participants who were greater than (>) 18 years of age and had confirmed diagnosis of psoriatic arthritis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time point.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1227
percentage of BSA
  Baseline (n=1227) | 9.7 (15.9)
  Change at Week 52 (n=796) | -6.6 (13.4)

3. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joints Count (DAS 28) at Week 52
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 100 mm; higher scores indicated greater affectation due to disease activity). DAS28 total score range: 0-10, where DAS28 less than or equal to (=<) 3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate disease activity and >5.1 = high disease activity.
Time Frame: Baseline, Week 52
Population: Efficacy analysis set included all participants who were >18 years of age and had confirmed diagnosis of psoriatic arthritis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1093
units on a scale
  Baseline (n=1093) | 4.8 (1.4)
  Change at Week 52 (n=629) | -2.2 (1.5)

4. Secondary Outcome: Change From Baseline in Ritchie Index at Week 52
Description: Ritchie index: the numerical measurement of joint tenderness (28 joints) in participants with arthritis. The number of quantitative evaluations of the pain experienced by the participants when the joints were subjected to firm pressure when exerted over the articular margin or in some instances by passive movement of the joint. Participant's reaction to pressure exerted by the physician were documented on 4-point scale, 0=not tender, 1=tender, 2=tender and caused wince, 3=reflexive effort to withdraw. Ritchie index was calculated as the total of the individual grades for all joints; ranged from 0 to 84, where higher score indicated higher tenderness.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1267
units on a scale
  Baseline (n=1267) | 9.9 (9.8)
  Change at Week 52 (n=851) | -4.1 (11.9)

5. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Week 52
Description: Physician global assessment of disease activity was measured on a 0 to 100 millimeter (mm) visual analog scale (VAS), with 0 mm = no disease activity to 100 mm = most possible disease activity.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1278
millimeter
  Baseline (n=1278) | 60.8 (18.8)
  Change at Week 52 (n=851) | -39.8 (24.2)

6. Secondary Outcome: Number of Participants With Nail Involvement
Description: Number of participants with psoriatic arthritis affecting the nails are reported.
Time Frame: Baseline, Week 12, 52
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1271
participants
  Baseline (n=1271) | 597
  Week 12 (n=1121) | 456
  Week 52 (n=837) | 259

7. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Week 52
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1124
milligram per deciliter (mg/dL)
  Baseline (n=1124) | 1.8 (3.0)
  Change at Week 52 (n=654) | -1.0 (3.0)

8. Secondary Outcome: Change From Baseline in Patient Assessment of Itching at Week 52
Description: Participants rated the severity of their psoriasis itching on a 0 (none) to 100 (most possible) scale.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1259
units on a scale
  Baseline (n=1259) | 36.8 (31.1)
  Change at Week 52 (n=838) | -22.7 (31.8)

9. Secondary Outcome: Change From Baseline in Patient Assessment of Pain at Week 52
Description: Participants rated the severity of their psoriatic arthritis-related pain on a 0 (none) to 100 (most possible) scale.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1276
units on a scale
  Baseline (n=1276) | 65.7 (21.6)
  Change at Week 52 (n=849) | -37.9 (28.3)

10. Secondary Outcome: Change From Baseline in 12-Item Short Form Health Survey (SF-12) at Week 52
Description: SF-12 questionnaire was used to determine participants' quality of life (QoL). It comprised 12 items which covered 8 concepts: physical functionality, role impairment due to physical problems, physical pain, perception of general health, vitality, social functionality, role impairment due to emotional problems, and psychological wellbeing. Results were presented in the form of 2 meta-scores, the physical component and the mental component, each ranged from 0 to 100. Higher scores=better QoL, positive changes from baseline=improvement in QoL.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1162
units on a scale
  Baseline: Physical component (n=1162) | 30.7 (8.5)
  Baseline: Mental component (n=1162) | 41.4 (11.7)
  Change at Week 52: Physical component (n=717) | 11.4 (10.8)
  Change at Week 52: Mental component (n=717) | 7.7 (12.3)

11. Other Pre Specified Outcome: Change From Baseline in Patient Global Assessment of Disease Activity at Week 52
Description: Measured using a 100 mm visual analog scale (VAS) ranging from 0 mm = very good to 100 mm = very bad.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1277
millimeter
  Baseline (n=1277) | 65.0 (20.6)
  Change at Week 52 (n=852) | -38.1 (27.3)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Participants With Psoriatic Arthritis
Serious Adverse Events (participants affected / at risk) | 77/1285
Other Adverse Events (participants affected / at risk) | 453/1285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Psoriatic Arthritis (N=1285)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Bradyarrhythmia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Cyanosis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Adrenal mass (Endocrine disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal wall disorder (Gastrointestinal disorders) | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Condition aggravated (General disorders) | 4
Drug ineffective (General disorders) | 1
Impaired healing (General disorders) | 1
Necrosis (General disorders) | 1
Nonspecific reaction (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Abscess limb (Infections and infestations) | 1
Abscess neck (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis Norwalk virus (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Liver function test abnormal (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Encephalitis (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Myelitis (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Alcohol rehabilitation (Surgical and medical procedures) | 1
Vascular operation (Surgical and medical procedures) | 1
Accelerated hypertension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphocele (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Psoriatic Arthritis (N=1285)
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Cardiac discomfort (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 1
Type IIb hyperlipidaemia (Congenital, familial and genetic disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 4
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Toxic nodular goitre (Endocrine disorders) | 1
Abnormal sensation in eye (Eye disorders) | 2
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 3
Conjunctivitis allergic (Eye disorders) | 1
Eye inflammation (Eye disorders) | 2
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 1
Iritis (Eye disorders) | 3
Keratitis (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Scleritis (Eye disorders) | 1
Sicca syndrome (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 18
Duodenal polyp (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Mucous stools (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Oral mucosal blistering (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 2
Stomach discomfort (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 4
Chills (General disorders) | 3
Condition aggravated (General disorders) | 41
Drug ineffective (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 20
Feeling cold (General disorders) | 1
Feeling hot (General disorders) | 1
General physical health deterioration (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site discolouration (General disorders) | 1
Injection site erythema (General disorders) | 66
Injection site hypersensitivity (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site inflammation (General disorders) | 2
Injection site irritation (General disorders) | 5
Injection site macule (General disorders) | 1
Injection site oedema (General disorders) | 2
Injection site pain (General disorders) | 2
Injection site papule (General disorders) | 1
Injection site pruritus (General disorders) | 32
Injection site rash (General disorders) | 6
Injection site reaction (General disorders) | 19
Injection site swelling (General disorders) | 16
Injection site urticaria (General disorders) | 2
Injection site warmth (General disorders) | 3
Local swelling (General disorders) | 1
Malaise (General disorders) | 2
Mucosal haemorrhage (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 2
Paradoxical pain (General disorders) | 1
Performance status decreased (General disorders) | 2
Pyrexia (General disorders) | 2
Sensation of foreign body (General disorders) | 2
Swelling (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Hepatocellular damage (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 5
Seasonal allergy (Immune system disorders) | 1
Type IV hypersensitivity reaction (Immune system disorders) | 1
Acute tonsillitis (Infections and infestations) | 2
Arthritis infective (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 19
Bronchopneumonia (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 2
Conjunctivitis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 3
Ear infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Febrile infection (Infections and infestations) | 4
Fungal skin infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Gastrointestinal infection (Infections and infestations) | 5
Helicobacter infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 2
Herpes virus infection (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 7
Infection in an immunocompromised host (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Laryngopharyngitis (Infections and infestations) | 1
Nail bed infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 50
Onychomycosis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 7
Oral infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Purulence (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 13
Rhinitis (Infections and infestations) | 2
Sinobronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 12
Skin infection (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Toxoplasmosis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 22
Urinary tract infection (Infections and infestations) | 10
Vaginal candidiasis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 3
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Forearm fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Antinuclear antibody increased (Investigations) | 1
Arthroscopy (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood pressure increased (Investigations) | 6
Body temperature increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 6
Haematocrit increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Liver function test abnormal (Investigations) | 8
Mean cell haemoglobin increased (Investigations) | 1
Mean cell volume increased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Transaminases increased (Investigations) | 5
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 2
White blood cell count decreased (Investigations) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 5
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2
Burning sensation (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Hyperaesthesia (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 3
Pseudoradicular syndrome (Nervous system disorders) | 1
Retrograde amnesia (Nervous system disorders) | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Trigeminal neuralgia (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Agitation (Psychiatric disorders) | 2
Alcoholism (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 9
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 10
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 17
Pruritus generalised (Skin and subcutaneous tissue disorders) | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 23
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 13
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Rosacea (Skin and subcutaneous tissue disorders) | 1
Scab (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4
Urticaria generalised (Skin and subcutaneous tissue disorders) | 1
Bone operation (Surgical and medical procedures) | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Dental operation (Surgical and medical procedures) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Intervertebral disc operation (Surgical and medical procedures) | 1
Joint injection (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Limb operation (Surgical and medical procedures) | 1
Meniscus operation (Surgical and medical procedures) | 1
Ossiculoplasty (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Results for Psoriasis Area and Severity Index (PASI) was not reported since it was not to be analyzed by rheumatologists as part of this study, as per planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.